CLINICAL TRIAL: NCT03260114
Title: Personal Activity Intelligence and Body Weight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2017/319/REK midt
Record Dates: First submitted 2017-08-23; First posted 2017-08-24 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Overweight; Obesity
Keywords: Physical activity; Body weight; Obesity
MeSH Terms: conditions — Overweight; Obesity; Motor Activity; Body Weight

STUDY DESIGN:
Intervention Model Description: We aim to recruit 30 persons who meet the eligibility criteria. Eligible participants will be randomized 1:1:1 to usual care (control group), to two different PAI eHealth Programs (PAI ≥ 100 and PAI = 50 to <100) (N = 10). To provide balance across the trial arms for sex, and age groups (<40, 40-55, >55 years), participants will be allocated remotely by concealed minimisation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Physical activity recommendations (No Intervention): Participants in this group will be advised to engage in physical activity recommendations from health authorities, i.e., 150 minutes per week of moderate intensity activity or 75 minutes per week of vigourous intensity activity or combination of both that results in same caloric expenditure.
- PAI equal to or more than 100 (Active Comparator): Participants in this group will be advised to obtain a PAI score of 100 or more over a week.
  Interventions: Other: Personal Activity Intelligence
- PAI between 50 and 99 (Active Comparator): Participants in this group will be advised to obtain a PAI score between 50-99 over a week.
  Interventions: Other: Personal Activity Intelligence

INTERVENTIONS:
Other: Personal Activity Intelligence — Participants randomized to the PAI eHealth program will be given a Mio Slice wristband (http://www.mioglobal.com/pai/), to measure the heart rate for calculating PAI. A weekly PAI of 100 can be achieved by a combination of different exercise intensities and the participants will, at any time, get information from the device (Mio Slice) (and the PAI App if they chose to use that as well) regarding how many minutes at specified heart rates is needed to achieve the weekly goal of 100 PAI. Participants will receive automatic feedback on a daily basis, and data will be automatically recorded on a secured server.
  Arms: PAI between 50 and 99; PAI equal to or more than 100

SUMMARY:
Physical activity is one of the key strategies used by public health agencies to combat the growing burden of obesity and non-communicable diseases. Adults around the world are recommended to engage in at least 150 minutes of moderate or 75 minutes of vigorous intensity activity per week, or a combination of moderate or vigorous activity that results in approximately the same total energy expenditure. However, majority of the population does not meet the physical activity recommendation. As barriers to physical activity, people mostly cite lack of time, self-motivation and confidence in the ability to be physically active. Cardiac Exercise Research Group (CERG) at Faculty of Medicine and Health Sciences at Norwegian University of Science and Technology recently developed Personal Activity Intelligence (PAI). PAI is a result of research based on the HUNT study where more than 60 000 individuals has been monitored over a period of more than 20 years. The goal is to make PAI the new world standard of activity tracking. PAI is an individual metric that makes sense of measured heart rate data, and significantly reduces the risk of lifestyle related diseases.

The purpose of the study is to obtain new knowledge about how the use of PAI is related to body weight.

DETAILED DESCRIPTION:
The prevalence of obesity in the Western world is continuously increasing and the amount of obese persons among the adult population in the United States is now 35%. As a result of this growing problem, it is important and necessary to find an efficient way to prevent further weight gain in the population.Physical activity is one of the key strategies used by public health agencies to combat the growing burden of non-communicable diseases. As a result adults around the world are recommended to engage in at least 150 minutes of moderate or 75 minutes of vigorous intensity activity per week, or a combination of moderate or vigorous activity that results in approximately the same total energy expenditure. However, majority of the population does not meet the physical activity recommendation. As barriers to physical activity, people mostly cite lack of time, self-motivation and confidence in the ability to be physically active.

Recently, using the HUNT study data, the Cardiac Exercise Research Group devised a simple metric termed Personal Activity Intelligence (PAI) which, using individual heart rate patterns of the body, estimates the optimal threshold of physical activity required for a specific objective: to decrease risk of premature death in an individual from the general population. The idea is to keep the weekly PAI score above 100. Since PAI is a personalized reflection of the body's response to physical activity based on heart rate, PAI score of 100 is specific to an individual. For example, a 100 PAI for a fit person is not the same as 100 PAI for an unfit person. PAI can be accumulated over a course of one week using physical activity of personal preference (i.e. walking, swimming, dancing, playing with grandchildren etc.) and allows for days with no activity as long as they are followed up by days of higher activity. However, the optimal amount and intensity (i.e. the number of PAI) of physical activity that would help for weight gain prevention still remains to be determined.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for clinical study is healthy participants with a BMI > 25 and < 40.

Exclusion Criteria:

We will exclude people with severe illness or disabilities that preclude or hinder completion of the study or make exercise contradicted, uncontrolled hypertension, arrhythmias or angina, participation in conflicting interventions, primary pulmonary hypertension, diagnosed dementia or chronic communicable infectious diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-08-24 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
changes in body weight - BMI | 12 weeks
  assessment of change in body weight/ BMI associated with PAI

SECONDARY OUTCOMES:
Cardiovascular Risk Factors | 12 weeks
  change in CVD risk factors associated with PAI

CONTACTS AND LOCATIONS:
Overall Officials: Javaid Nauman, PhD, Principal Investigator — Norwegian University of Science and Technology, Trondheim, Norway
Locations (1):
- St. Olav´s University Hospital, Trondheim, Sor Trondelag, Norway

IPD SHARING:
Plan to Share IPD: Undecided